CLINICAL TRIAL: NCT04532359
Title: STABICAN : Measurement of Implant Stability by Analysis of the Resonance Frequency in Patients Treated for Cancer of the Upper Aero-digestive Tract
Brief Title: Measurement of Implant Stability by Resonance Frequency Analysis in Patients Treated for an Upper Aero-digestive Tract Cancer
Acronym: STABICAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: STABICAN - ET20-099
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Cancer
Keywords: Upper aero-digestive tract Cancer; Dental implant placement
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Implant placement — Implant placement

SUMMARY:
The primary objective is to describe the evolution of implant stability between the date of implant placement and 3 months later when the implant is implementated in patients treated for cancer of the upper aero-digestive tract

DETAILED DESCRIPTION:
Oral implantology is widely used during prosthetic rehabilitation in healthy patients but also in patients presenting cancers of the upper aero-digestive tract.

Systems for measuring implant stability using resonance frequency analysis exist and are used clinically by some practitioners, such as the Ostell® system from W&H. These systems make it possible to determine the osseointegration of the implant, and thus the appropriate time to insert the implant, by comparing the value obtained with average values.

Implant survival rates are lower for implants placed in irradiated bone, with an implant stability quotient value identical to implant placement but lower after osseointegration. Only one study shows implant stability quotient values> 60 with a success rate of 100% at 41 months on implants placed in patients having received radiotherapy. However, no clinical study has investigated the kinetics of osseointegration and the stability of implants placed on a microanastomosis fibula flap as part of aesthetic and prosthetic reconstruction after cancer of the upper aero-digestive tract.

ELIGIBILITY:
Inclusion Criteria:

* Patient with squamous cell carcinoma of the upper aero-digestive tract (oral cavity, oropharynx, hypopharynx
* Patient having been treated by external radiotherapy and/or having benefited from a microanastomosis fibula flap
* Patient going to undergo a surgical intervention with placement of dental implant(s) in an irradiated area or in the microanastomosis fibula flap
* Non-opposition to the study

Exclusion Criteria:

* Patient having difficulties speaking and understanding French
* Patient under tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with squamous cell carcinoma of the upper aero-digestive tract (oral cavity, oropharynx, hypopharynx) who are going to undergo a surgical intervention with placement of dental implant(s) in an irradiated area or in the microanastomosis fibula flap.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of implant stability in patients treated for cancer of the upper aero-digestive tract between placement and 3 months after placement | At 3 months after implant placement
  Measure with Osstell Beacon device (Implant Stability Quotient : value from 1 to 100)

SECONDARY OUTCOMES:
Evaluation of the association between the type of bone (maxilla/mandible and fibula) and implant stability | At 3 months after implant placement
  Correlation between the type of bone (maxilla / mandible and fibula) and implant stability
Evaluation of the correlation between the irradiation dose received at the implant site and implant stability | At 3 months after implant placement
  Correlation between the irradiation dose received at the implant site and implant stability

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Gaëlle CHAUX-BODARD, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France